CLINICAL TRIAL: NCT06009354
Title: Effectiveness of Multi-Component Training in Lower Extremity Release Surgery
Brief Title: Effectiveness of Education in Relaxation Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP gevşetme
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The study group will receive multi-component training in addition to the usual practices. In the multi-component training content, self-massage applications performed by the patient's relatives, joint range of motion applications for the extremities, respiratory training, issues to be considered in activities of daily living, training on the use of assistive devices and training on methods of coping with pain kinesiophobia will be given to the patient's relatives through a video.
  Interventions: Other: Rehabilitation
- Control Group (Active Comparator): The control group will receive the usual post-operative applications (elevation, rest, cold application, stretching).
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — The control group will receive post-operative usual practices. The study group will receive multi-component education in addition to the usual practices.

SUMMARY:
The study will be carried out with volunteer patients who are followed up by the Orthopedics and Traumatology outpatient clinic of Muğla Training and Research Hospital and diagnosed with Cerebral Palsy and meet the study criteria. The evaluations will be performed in the Orthopedics and Traumatology outpatient clinic of Muğla Training and Research Hospital. This study was planned to investigate the effectiveness of multicomponent home activities and family child education against conventional postoperative practices in children with CP who underwent lower extremity tendon release surgery. Objective functional status, spasticity levels, pain levels, kinesiophobia levels and gait quality of the patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children with walking CP between the ages of 4-18 years who have undergone lower extremity orthopedic surgery and at least 2 months have passed (leaving the acute and subacute period behind)
* Gross Motor Function Classification (GMFCS) level 1 (walks without restrictions), 2 (walks with restrictions) or 3 (walks using hand-held mobility aids)
* Understand simple commands
* Signing the consent form

Exclusion Criteria:

* Circumstances that would interfere with conducting assessments or communicating
* Lack of cooperation during the study
* Presence of severe mental retardation
* Presence of botulinum toxin application in the last 6 months

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK) | Change from Baseline TSK at 8 weeks
  The questionnaire is a 17-item scale developed to measure fear of movement/reinjury. The normal score range is between 17 and 68.
Pain Catastrophising Scale (PCS) | Change from Baseline PCS at 8 weeks
  Scale is used to assess the patient's feelings and thoughts about pain and disaster. The total score ranges from 0 to 52 points. A high score indicates a bad situation.
Timed Up and Go Test (TUG) | Change from Baseline TUG at 8 weeks
  Participants sit in a chair with arms, hips and knees bent approximately 90◦ and feet resting on the floor. Lower limb orthoses are worn if used. Participants are asked to stand up, walk 10 steps, walk around a mark on the floor, walk back to the chair and sit down. The timing of the TUG test starts with the standing movement after the "ready, go" signal and ends when the participants are seated in the chair and the movement is finished.
One Leg Standing Test (OLST) | Change from Baseline OLST at 8 weeks
  Children are tested standing on one leg using their right and left leg respectively. The test is repeated on a hard surface with eyes open and closed. The child is asked to place both hands on the hips and look at a target on the wall at eye level at a distance of 1 meter. The child is asked to stand with one leg while keeping the other leg in a 90 degree flexion position. A stopwatch is used to record the time the child can hold the test position. The examiner ends the test if the child can hold the position for more than 30 seconds and records the elapsed time.
Functional Reach Test (FRT) | Change from Baseline FRT at 8 weeks
  The subject stands sideways next to a wall and flexes the shoulder 90 degrees. The 3rd metacarpal level is marked on the wall. The subject reaches as far as he/she can without taking a step. The 3rd metacarpal line is marked again. The difference between the marks is measured and noted.
Gross Motor Function Classification System (GMFCS) | Change from Baseline GMFCS at 8 weeks
  The aim of this classification system is to provide a standardized classification of motor disability patterns in children with CP. It is a five-level ordinal grading system for classifying gross motor function in a child with CP, with level I representing the least limitation and level V the most limitation. At level I, children show mild involvement and can perform most of the activities of their peers. At level V, children show severe involvement, lacking head control and sitting balance.
Modified Ashworth Scale (MAS) | Change from Baseline MAS at 8 weeks
  The Modified Ashworth Scale (MAS) is an indirect measure of the nature of spasticity. The MAS is a scale of perceived resistance (tone) to passive movement of the limb and is an adaptation of the original Ashworth Scale with the addition of the 1+ category.
Wong-Baker FACES Pain Rating Scale (WBFPRS) | Change from Baseline WBFPRS at 8 weeks
  The Wong-Baker FACES Pain Rating Scale shows six faces with increasing degrees of pain from left to right and each face is rated out of 10. 0 indicates no pain, 2 indicates a little pain, 4 indicates a little more pain, 6 indicates more pain, 8 indicates a lot of pain, and 10 indicates the worst pain.
FLACC Behavioral Pain Assessment scale | Change from Baseline FLACC at 8 weeks
  The FLACC scale scores pain intensity by rating five behaviors (face, legs, activity, consolability and crying) to obtain a score out of 10. The FLACC scale is a composite of five behaviours ('face', 'legs', 'activity', 'cry' and 'consolability') considered indicative of pain that can be detected and graded by an observer. Each item is scored on a zero to two scale resulting in a pain intensity score ranging from zero to 10. The original instructions for use recommended observing the child for one to five minutes and matching the observed behaviours to those described in the scale for each item.
Wisconsin Gait Scale (WGS) | Change from Baseline WGS at 8 weeks
  The WGS, consisting of four subscales, evaluates 14 gait parameters which can be observed in the affected leg during consecutive gait stages, i.e. stance, toe off, swing and heel strike phases. Additionally, it accounts for the use of hand held gait aid while walking. The first subscale is designed to assess spatiotemporal gait parameters, while kinematic parameters are evaluated by subscale one, two, three and four. In all the items of the scale subjects can score from 1 to 3 points, except for Item One (1-5 points) and Item Eleven (1-4 points). The total number of points falls between 13.35 and 42, a higher score corresponding to greater gait impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, PhD, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No